CLINICAL TRIAL: NCT06638242
Title: Indicators of Quality Care and Services for Adults With Acute Ischemic Stroke in Different Types of Hospitals in Quebec (IndiQ-AVC) : Research Protocol
Brief Title: Indicators of Quality Care and Services for Adults With Acute Ischemic Stroke in Different Types of Hospitals in Quebec : Research Protocol
Acronym: IndiQ-AVC
Status: Completed | Type: Observational
Sponsor: Amelie Belanger (Other)
Responsible Party: Sponsor-Investigator, Amelie Belanger, Assistant professor, department of nursing, Université du Québec à Trois-Rivières
Organization: Université du Québec à Trois-Rivières (Other)
Other Study IDs: MP-29-2022-606
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Stroke
Keywords: clinical and organizational quality incdicators; practices assessment; stroke acute phase; interdisciplinarity
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to describe the performance of care and services offered to people hospitalized with ischemic stroke. More specifically, this study aims to answer the following questions:

* Is stroke care and service delivered to the population optimally?
* Are these services equitable, regardless of the hospital where the patient is hospitalized?
* Are all patients treated in the same way, regardless of individual characteristics such as age, sex or risk factors?

An evaluation of the quality of practices will be carried out on the health records of patients hospitalized in different hospital centers in Quebec such as a subspecialized center, a regional center and a center in a remote region. An in-depth analysis will also be conducted to determine whether certain individual patient characteristics may influence how they are managed during a stroke.

ELIGIBILITY:
Inclusion Criteria:

- Adults 18 years old or over with ischemic stroke requiring hospitalization in an acute care unit or special stroke unit

Exclusion Criteria:

* Adults with hemorrhagic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with ischemic stroke All persons hospitalized for ischemic stroke within the 6 months preceding approval of the Research Ethics Board (REB). The study will be conducted based on their health records.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Descriptives analyses | All persons hospitalized for ischemic stroke within the 6 months preceding approval of the Research Ethics Board (REB).
  Descriptive analyses will be completed to assess clinical and organizational practices in hospital centers from patients'health records

CONTACTS AND LOCATIONS:
Locations (1):
- Centre intégré universitaire de santé et services sociaux de la Mauricie et du Centre-du-Québec, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT06638242/Prot_000.pdf